CLINICAL TRIAL: NCT03805815
Title: Development of Diagnosis Algorism for Paroxysmal Arrhythmia Using Ultra-thin Resistive Membrane: a Pilot Study
Brief Title: Clinical Implication of the Tunable Crack Sensor
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Professor of Medicine / Cardiology, Seoul National University Hospital
Other Study IDs: H-1808-177-969
Record Dates: First submitted 2018-12-30; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Blood Pressure
Keywords: blood pressure; crack sensor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: tunable crack sensor — blood pressure monitoring via crack sensor

SUMMARY:
[Development of diagnosis algorism for paroxysmal arrhythmia using ultra-thin resistive membrane: a pilot study] Comparison of blood pressure via tunable crack sensor and invasive pressure wire

DETAILED DESCRIPTION:
To develop a diagnosis algorism for paroxysmal arrhythmia using ultra-thin resistive membrane, we will compare the blood pressure measured via a tunable crack sensor and that measured by a invasive pressure wire

ELIGIBILITY:
Inclusion Criteria:

A case of suspected coronary artery disease at Seoul National University Hospital for the purpose of coronary angiography

* At least 19 years old
* If he/she hears enough explanation about clinical research and intends to participate in clinical research himself

Exclusion Criteria:

* Under 19 years old
* Refusal to participate in clinical studies
* If the cognitive function is weak enough not to understand the explanation of the clinical study and to make voluntary decisions accordingly

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A case of suspected coronary artery disease for the purpose of coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Blood pressure monitoring using tunable crack sensor | immediately
  Systolic blood pressure and diastolic blood pressure by using tunable crack sensor

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul national university hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kang D, Pikhitsa PV, Choi YW, Lee C, Shin SS, Piao L, Park B, Suh KY, Kim TI, Choi M. Ultrasensitive mechanical crack-based sensor inspired by the spider sensory system. Nature. 2014 Dec 11;516(7530):222-6. doi: 10.1038/nature14002. PMID 25503234